CLINICAL TRIAL: NCT04332393
Title: The Effect of Metformin in Pregnant Women Who Received Antenatal Corticosteroids on Glycemic Control and the Rate of Neonatal Hypoglycemia - Multicenter Prospective Randomized, Controlled Trial
Brief Title: Metformin to Treat Corticosteroids-induced Hyperglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-20POR
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Preterm; Glycemic Control; Corticosteroids Induced Hyperglycemia
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin group (Experimental)
  Interventions: Drug: Metformin
- No treatment group (No Intervention)

INTERVENTIONS:
Drug: Metformin — Metformin tablets according to glycemic control. Initial dose: 425 mg before meals (breakfast, lunch and supper) and 1700 mg around 22:00. Modifications may take place according to glycemic control
  Arms: metformin group

SUMMARY:
Antenatal corticosteroids, particularly, betamethasone is routinely administered to pregnant women at risk for preterm delivery to improve neonatal outcomes.

Although antenatal betamethasone was shown to induce both maternal hyperglycemia and neonatal hypoglycemia, to date, there is insufficient data to establish whether treatment for maternal hyperglycemia, particularly, metformin, will decrease the risk for neonatal hypoglycemia, particularly of preterm neonates.

In the present study the investigators will examine the effect of treatment with metformin on maternal glycemic control and hypoglycemia in preterm neonates following maternal betamethasone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving betamethasone from 24 to 36.5 gestational weeks
* Before or within 24 hours following the first dose of betamethasone
* ≥18 years old

Exclusion Criteria:

* Women with pre-gestational and gestational diabetes mellitus (GDM)
* Known allergic sensitivity to metformin
* Known chronic heart failure
* Known chronic renal failure
* Refuse to participate
* Refuse to perform glucose challenge test/glucose tolerance test later on

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Mean maternal daily glucose values | Up to 4 days
  According to daily glucose charts
The rate of neonatal hypoglycemia in preterm deliveries (<37 gestational weeks) | Up to 7 days after delivery or discharge (which ever comes first)

SECONDARY OUTCOMES:
Mean maternal daily pre-prandial glucose values | Up to 4 days
  According to daily glucose charts
Mean maternal daily post-prandial glucose values | Up to 4 days
  According to daily glucose charts
Percent of abnormal values in the daily glucose chart | Up to 4 days
  According to daily glucose charts
Rate of cesarean sections and operative deliveries | At delivery
Rate of neonates who will be admitted to the neonatal intensive care unit | Up to a week after delivery
  APGAR scale of 0-worst and 10-best
Apgar score at 1 and 5 minutes | At delivery
Cord blood pH levels (when taken) | At delivery
The rate of neonates with hyperbilirubinemia | Up to 7 days after delivery or discharge (which ever comes first)
Neonatal mean head circumference | Up to 7 days after delivery or discharge (which ever comes first)
Neonatal mean birth weight | at delivery
The rate of fetal malformations and developmental disorders | Up to 7 days after delivery or discharge (which ever comes first)
Mean and lowest neonatal blood glucose values in preterm neonates | Up to 7 days after delivery or discharge (which ever comes first)
The rate of maternal adverse effects | 48 hours

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Baruch Padeh Medical center, Poriya, Tiberias, North
  - Emek medical center, Afula
  - Galilee medical center, Nahariya
  - Ziv medical center, Safed

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared according to the local review board regulations

REFERENCES:
- [Derived] Yefet E, Massalha M, Talmon G, Labay A, Matanis M, Sleman E, Nassra R, Frank Wolf M, Sgayer I, Lowenstein L, Nachum Z. Metformin, Maternal Glycemic Control, and Neonatal Hypoglycemia After Antenatal Steroids: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2552807. doi: 10.1001/jamanetworkopen.2025.52807. PMID 41511771